CLINICAL TRIAL: NCT01185756
Title: Can we Better Select Patients With Heart Failure for a Primary Prevention Indication of Implantable Cardioverter Defibrillator (ICD)? Evaluation of the Diagnostic Value of 123I Meta-iodobenzylguanidine (MIBG)
Brief Title: MIBG Scintigraphy as a Tool for Selecting Patients Requiring Implantable Cardioverter Defibrillator (ICD)
Acronym: MISTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM : 08085
Record Dates: First submitted 2010-07-09; First posted 2010-08-20 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure; Sudden Death
Keywords: Heart failure; Sudden death; Implantable Cardioverter Defibrillator; MIBG scintigraphy
MeSH Terms: conditions — Heart Failure; Death, Sudden | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICD implantation (Experimental): MIBG for diagnostic purpose:
  MIBG scintigraphy for diagnostic purpose
  Interventions: Radiation: MIBG for diagnostic purpose

INTERVENTIONS:
Radiation: MIBG for diagnostic purpose — All patients will undergo the diagnostic test specific to the study.

SUMMARY:
The aim of the study is to assess the cardiac innervation in patients with heart failure to better select candidates for an implantable cardioverter defibrillator. Cardiac innervation will be assessed using an imaging agent administered intravenously.

DETAILED DESCRIPTION:
The survival benefit provided by implantable cardioverter defibrillator (ICD) for primary prevention of sudden cardiac death in heart failure compared to medical treatment alone is well established. First limited to the most severe patients, the indications have gradually been extended in accordance with the results of more recent studies. This beneficial effect in terms of public health is accompanied by an increase in health spending which threatens to grow strongly at short and medium term. However, the majority of ICDs implanted will not be solicited because of the overall low incidence of severe ventricular arrhythmias in the population meeting the implantation criteria. To optimize our resources, it is therefore important to better assess the risk of sudden death in those patients candidates for ICD implantation.

The overactivation of NEURO-humoral systems plays an important role in the progression of heart failure, and in the occurrence of ventricular arrhythmias. The iodine-123 meta-iodobenzylguanidine scintigraphy (MIBG), is a functional imaging method that can noninvasively evaluate cardiac sympathetic innervation. It has been shown that cardiac adrenergic hyperactivation estimated by MIBG scintigraphy was associated with a poor outcome, and that its value was independent and superior to other prognostic factors in heart failure. More importantly, the risk of occurrence of major cardiac events is minimal when the cardiac uptake of MIBG is high. Furthermore, plasma natriuretic peptides (particularly BNP and NT-proBNP), which are other indicators of the NEURO-hormonal activation used in the diagnosis and assessment of prognosis in heart failure, are predictive of the risk of occurrence of sudden death in the same population. In summary, the MIBG scintigraphy and NT-proBNP are two prognostic markers in heart failure related to the degree of NEURO-hormonal dysfunction, and have a good negative predictive value of mortality. Their combined use could therefore help identify patients at low risk of severe arrhythmias.These tests are not currently part of heart failure diagnosis in patients who are candidates for ICD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ICD in primary prevention according to European Society of Cardiology guidelines

Exclusion Criteria:

* Secondary prevention indication of ICD
* Acute coronary syndrome within the last 40 days
* Revascularization procedure (bypass or percutaneous coronary angioplasty) performed within the last 3 months of planned
* Pregnancy or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the cardiac MIBG uptake ratio for identification of patients at very low risk of severe ventricular arrhythmias. | 1-3 months
  Description appropriate therapy delivered by the ICD, or sustained ventricular tachycardia.

SECONDARY OUTCOMES:
Sudden cardiac death | 1-3 months
Overall mortality | 1-3 months
Assessment of the cardiac MIBG uptake ratio for identification of patients at very low risk of severe ventricular arrhythmias. | every 6 months during 3 years
  description appropriate therapy delivered by the ICD or sustained ventricular tachycardia
sudden cardiac death | every 6 months during 3 years
Overall mortality | every 6 months during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Le Guludec, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided